CLINICAL TRIAL: NCT05921682
Title: Early Body Temperature Targets and Relationship With Prognosis in Patients With Heat Stroke
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Yiwu Central Hospital (Other); Jinhua People's Hospital (Other); Jinhua Municipal Central Hospital (Other); Dongyang People's Hospital (Other); Lanxi People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0517
Record Dates: First submitted 2023-05-23; First posted 2023-06-27 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Heat Stroke
Keywords: heat stroke, body temperature, outcomes
MeSH Terms: conditions — Heat Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with heat stroke: Patients with heat stroke presenting to the emergency department at the study site
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — This study is an observational study. Patients will receive conventional cooling measures and organ function support.

SUMMARY:
The goal of this observational study is to explore the optimal target body temperature in first 24 hours and the relationship between body temperature and adverse outcomes of heat stroke.

The main questions it aims to answer are:

* the optimal target body temperature at 0.5 h, 2 h, and the lowest body temperature of heat stroke.
* the best body temperature at the cutting point of stop cooling.
* The relationship between the volume and speed of ice saline infusion and the cooling effect.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years; ② diagnosed as heat stroke; ③ Informed consent from patients or family members.

Exclusion Criteria:

* need immediate cardiopulmonary resuscitation; ② transferred from another hospital; ③ with severe underlying organ insufficiency; ④ pregnant women.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Comprehensive tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-28 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
mortality | up to 90 days
  Number of participants who dead during hospitalization
organ damage | up to 90 days
  Number of participants with organ damage, including but not limited to brain, lung, heart, kidney, liver and coagulation

SECONDARY OUTCOMES:
continuous renal replacement therapy | up to 90 days
  Number of participants who need CRRT
length of ICU stay | up to 90 days
  The length patient stay in ICU
length of hospital stay | up to 90 days
  The length patient stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Lan Chen, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (6):
- China (6):
  - Yiwu Central Hospital, Yiwu, Zhejiang
  - Dongyang People's Hospital, Dongyang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Jinhua Municipal Central Hospital, Jinhua
  - Jinhua People's Hospital, Jinhua
  - Lanxi People's Hospital, Lanxi